CLINICAL TRIAL: NCT02857985
Title: Evaluation of Infarct Size With 3D Rotational Angiography
Acronym: EVATIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-749
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; MRI; rotational angiography
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with Myocardial Infarction (Experimental)
  Interventions: Device: 3D RA; Device: MRI

INTERVENTIONS:
Device: 3D RA — 3D RA is realised just after angioplasty.
Device: MRI — MRI is realised between 24h and 96h post angioplasty.

SUMMARY:
The size of the infarct is particularly important prognostic marker. It is clearly established that the extent of the infarct is not only correlated to mortality, but also long-term adverse events. The evaluation of the infarct size at the acute phase of the disease is therefore an essential clinical tool to adapt the immediate treatment and follow-up of patients. It is therefore crucial to have techniques that are effective, precise, reproducible, and easily performed during the acute phase to quantify the size of the infarct following angioplasty. Myocardial scintigraphy and cardiac MRI have been the standard examinations for the evaluation of infarct size. However, these exams are difficult to perform during the acute phase of the infarct owing to difficulties in monitoring unstable patients and the limited availability of the apparatus. It is for this reason that the investigators would like to investigate the rotational angiography (RA), which is comparable to a scanner in its mode of action but does not require transfer of patients as performed using the same apparatus that used for diagnostic coronarography and therapeutic angioplasty. RA is a radiological technique that uses the system employed for coronagraph, and consists rotating the fixed C-Arm around the patient and acquisition of a series of images that are then reconstituted. The investigators propose to evaluate the size of the infarct using RA in comparison with cardiac MRI (standard examination) performed as soon as possible after RA and the investigators hope to demonstrated that RA allows the measurement of an infarct as precisely as cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for myocardial infarction and fulfilling the following criteria:

  * Transitory or persistent ST elevation
  * Coronary occlusion (TIMI 0) treated by angioplasty or thrombotic acute stenosis treated or not by angioplasty
* Planned coronarography
* With social security coverage
* Not under any legal protection;
* The consent form signed.

Exclusion Criteria:

* Patient unconscious or confused;
* Presenting:

  * cardiogenic shock;
  * or signs of cardiac insufficiency;
  * or sustained cardiac arrhythmia;
  * or atrial fibrillation;
  * or sustained extrasystole;
  * or high degree block;
* Contraindication for MRI;
* Known history of hypersensitivity to MRI contrast agent;
* Risk of pregnancy or proven pregnancy based on interview data;
* Breast feeding;
* Patient subject to legal guardianship by a court;
* Incapacity to express consent;
* Patient not or badly understanding French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03-09 (Actual); Primary Completion 2013-09-07 (Actual); Study Completion 2013-09-07 (Actual)

PRIMARY OUTCOMES:
infarct size measured by RA | Day 1
infarct size measured by MRI | Day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No